CLINICAL TRIAL: NCT05025410
Title: General Anesthesia Using Remimazolam and Remifentanil Without Neuromuscular Blocking Agent: Prospective Observational Study
Brief Title: Remimazolam and Remifentanil Without Neuromuscular Blocking Agent
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Principal investigator, Seoul National University Bundang Hospital
Other Study IDs: B-2109-706-301
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Myoma;Uterus; Polyp Endometrium; Unspecified Condition Associated With Female Genital Organs and Menstrual Cycle
MeSH Terms: conditions — Myofibroma | interventions — remimazolam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General anesthesia using remimazolam and remifentanil: Adult female patients scheduled for gynecological surgery under general anesthesia using remimazolam and remifentanil
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Loading for anesthesia induction: Remimazolam 6 mg/kg/h until loss of consciousness Continuous infusion for anesthesia maintenance: Remimazolam 1-2 mg/kg/h under the Bispectral index monitoring

SUMMARY:
Remimazolam is a novel drug approved for induction and maintenance of general anesthesia. This study aims to check the appropriate dose and patient response by administering remimazolam and remifentanil in surgery that does not require a neuromuscular blocking agents.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman scheduled for gynecological surgery under general anesthesia
* American Society of Anesthesiology grade 1 or 2
* When using a laryngeal mask airway to maintain general anesthesia

Exclusion Criteria:

* Underlying diseases: liver, kidney, brain nervous system, glaucoma
* Patients with BMI greater than 30 and less than 18.5
* Patients diagnosed with sleep apnea
* Alcohol or drug dependent patients
* Patients with severe or acute respiratory failure
* Lactose intolerance
* Dextran 40 hypersensitivity
* Patients in shock or coma

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult woman scheduled for gynecological surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Remimazolam induction dose | During the anesthesia induction (from initiation of anesthesia until the insertion of laryngeal mask airway)
Remimazolam maintenance dose | During the anesthesia maintenance (from the insertion of laryngeal mask airway until stopping remimazolam infusion)

SECONDARY OUTCOMES:
Use of rescue midazolam | During the anesthesia (from initiation of anesthesia until stopping remimazolam infusion)
Use of rescue rocuronium | During the anesthesia (from initiation of anesthesia until stopping remimazolam infusion)
Use of flumazenil | During the anesthesia recovery (from stopping remimazolam infusion until the recovery of consciousness)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park I, Cho M, Nam SW, Hwang JW, Do SH, Na HS. Total intravenous anesthesia induced and maintained by a combination of remimazolam and remifentanil without a neuromuscular blocking agent: a prospective, observational pilot study. BMC Anesthesiol. 2022 Jul 26;22(1):237. doi: 10.1186/s12871-022-01779-2. PMID 35883039